CLINICAL TRIAL: NCT05096494
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Study to Evaluate the Safety and Efficacy of SP-103 in Subjects With Moderate to Severe Acute Lower Back Pain
Brief Title: Safety and Efficacy of SP-103 in Subjects With Moderate to Severe Acute Lower Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-103-02
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Moderate to Severe Acute Lower Back Pain
Keywords: lbp; lower back pain; lidocaine; topical system; patch
MeSH Terms: conditions — Hypotension; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-103 (Experimental): One SP-103 transdermal system is worn 12 hours per day for 28 days on the lower back.
  Interventions: Drug: SP-103
- Placebo (Placebo Comparator): One placebo transdermal system is worn for 12 hours per day for 28 days on the lower back
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-103 — SP-103 topical system is worn daily for 12 hours per day for 28 days
  Arms: SP-103
Drug: Placebo — Placebo topical system is worn daily for 12 hours per day, for 28 days
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel group, multicenter study to evaluate the safety and efficacy of SP-103 in subjects with moderate to severe acute lower back pain.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel group, multicenter study to evaluate the safety and efficacy of SP-103 in subjects with moderate to severe acute lower back pain. Three to 7 days after the Screening Visit, subjects will return for a Baseline visit to verify electronic Diary compliance, collect urine samples for a drug screen and pregnancy test (for women of child-bearing potential), and complete baseline clinical rating scales.

If subjects meet all the study inclusion criteria and none of the exclusion criteria, subjects will be randomized into the study. Subjects are expected to apply investigational product for 12 hours per study day) study days 1 through 28 and to record the time of investigational product applications and removals an electronic diary.

Subjects will capture daily numeric pain rating scores and topical adhesions assessments in the electronic diary each evening prior the removal of investigational product.

On day 28, subjects will return to the study site to complete the End of Study visit.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, write, and understand the informed consent prior to beginning any study procedures.
* Male or female, age 18 to 75 years (inclusive).
* Based on medical history, current episode of lower back pain (LBP) must have been present for not more than 3 months.
* Currently experiencing localized area of muscular tenderness in lower back area between the lowest rib and the gluteal fold in moderate-to-severe intensity as evaluated by the investigator.
* If deemed necessary by the Investigator, has a willing partner (facilitator) that can apply study drug to the designated anatomical area.
* Intact skin at the site of pain with no skin breakdown or inflammation.
* Negative urine drug screen.
* Average LBP numeric pain rating scale (NPRS) score of sufficient severity over the last 24 hours.
* Sufficiently compliant with electronic Diary entries.
* If a woman of childbearing potential (WOCBP) agrees to use an effective method of birth control during the study.
* If a WOCBP (i.e., not surgically sterile or at least 2 years postmenopausal), must have negative pregnancy tests.
* Have the means and willing to conduct a video-based televisits.
* Reviewed all study specific educational materials and has, in the opinion of the Investigator, the cognitive abilities to understand and appropriately complete all study mandated procedures.

Exclusion Criteria:

* A body mass index (BMI) ≥40 kg/m2
* Significant pain unrelated to LBP which, in the Investigator's and/or Sponsor's opinion, would significantly compromise assessment of LBP.
* Duration of current LBP episode greater than 3 months.
* Has LBP due to any of the following pathologies: infection, neoplasia, severe metabolic or structural disease of spine, lumbar radiculopathy, osteoporosis, hip dysplasia, inflammatory arthritis, ankylosing spondylitis, Paget's disease, cauda equina syndrome, gout, pseudogout, fibromyalgia, active post surgical pain, or pain over neurostimulator battery site.
* Has LBP caused by major trauma.
* Has had history of lower back surgery.
* Has excess hair that cannot be clipped (shaving/waxing is not permitted to the area), excess tattoo(s), or other dermatological conditions in the topical system application area that may interfere, in the opinion of the Investigator, with administration, efficacy, and safety evaluations.
* Use of Qutenza on the back within 3 months.
* Use of opioids for ≥4 days per week.
* Unwilling to discontinue all opioids, NSAIDs, other analgesics, or non-pharmacological therapy intended to treat LBP such as tapes (e.g., KT tape®), heated heat therapy (e.g., heat packs/pads, sauna, hot tub), or cold therapy (e.g., ice pack) for the duration of the trial.
* Unwilling to maintain the same regimen of physical activities throughout study participation.
* Anxiety or depression based on the Hospital Anxiety and Depression Scale scores, or has a major psychiatric disorder not controlled with medication that would interfere with clinical pain scores or participation in the trial.
* Alcohol dependence, illicit drug use based on urine screen (including recreational or medical use of tetrahydrocannabinol (THC) -containing substances, or non-prescribed use of controlled drug substances), or drug addiction.
* Current COVID-19 infection, if tested according to local requirements.
* Clinically significant abnormalities which, in the opinion of the Investigator, may compromise subject safety.
* Significant motor impairment, sensory deficits, pain in lower extremities, and/or new onset of bowel/bladder impairment based on history and neurological examination.
* History of fibromyalgia or diagnosis of fibromyalgia based on American College of Rheumatology 2016 criteria.
* History of malignancy or evidence of malignancy, lymphoproliferative, or neoplastic disease except for successfully treated basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia within 5 years.
* If female, is lactating/breastfeeding, plans to breastfeed, or plans to become pregnant while participating in the study.
* Known history of any clinically significant or unstable medical condition, any other disorder, condition or circumstance (including secondary gain) which in the opinion of the Investigator has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.
* Has a serious illness that resulted in recent hospitalization.
* History of Myocardial Infarction within the last 6 months, New York Heart Association Class III or higher congestive heart failure, and any clinically significant ECG abnormality or arrhythmias.
* Has a hypersensitivity or allergy to the investigational compound/compound class being used in this study or any ingredients of this medication, including but not limited to lidocaine and amide compounds.
* Use of opioid and non-opioid analgesics for indications other than back pain.
* Use of any investigational drug and/or device within 28 days or is scheduled to receive an investigational drug other than blinded study drug while participating in the study.
* Involvement in an ongoing or planned worker's compensation claim, disability claim, or litigation related to any pain problem, receiving payments for a settled claim, awaiting pending payment for a settled claim, or any additional secondary gain in the opinion of the Investigator.
* Is an employee, family member, or student of the Investigator or clinical site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 days
Numeric Pain Rating Scale (0-10, 0 is no pain, 10 is worst pain imaginable) | 7 days

SECONDARY OUTCOMES:
Oswestry Disability Index (0-100, 0 is with no disability, 100 is the maximum disability) | Day 7 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, Study Director — Chief Medical Officer
Locations (10):
- United States (10):
  - Arizona Research Center, Phoenix, Arizona
  - Costal Clinical Research Specialists, Fernandina Beach, Florida
  - Costal Clinical Research Specialists, Jacksonville, Florida
  - Horizon Clinical Research, Newnan, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Anaesthesia Research Specialists, Chicago, Illinois
  - Neuroscience Research Center, Overland Park, Kansas
  - Neuroscience Institute, Overlook Medical Center, Summit, New Jersey
  - Western Reserve Hospital, Cuyahoga Falls, Ohio
  - Scilex Research Site 08, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No